CLINICAL TRIAL: NCT04561258
Title: Phase 1 Study to Evaluate the Safety of Genetically Modified, Autologous T Cells in Participants With HIV That is Well-Controlled on Antiretroviral Therapy
Brief Title: Study to Evaluate the Safety of a Gene and Cell Therapy Product in Participants With HIV That is Well-Controlled on Antiretroviral Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Gene Technologies International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGT-HC168
Record Dates: First submitted 2020-09-14; First posted 2020-09-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Cohort (Experimental): A single infusion of ≥1x10e8 and <1x10e9 genetically modified T cells.
  Interventions: Biological: AGT103-T
- High Dose Cohort (Experimental): A single infusion of ≥1x10e9 and <5x10e9 genetically modified T cells.
  Interventions: Biological: AGT103-T

INTERVENTIONS:
Biological: AGT103-T — An autologous, genetically modified PBMC product enriched with HIV-specific and resistant CD4 T cells

SUMMARY:
This is a Phase 1 study to assess the safety of a gene and cell therapy for autologous donor lymphocyte infusion in HIV+ participants with well-controlled viremia on antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18-60 years
2. Documented HIV infection for ≥3 years
3. Suppression of HIV to <50 copies of viral RNA/mL plasma for ≥2 years. Participants who had intermittent, isolated episodes of detectable low-level viremia (<500c/mL; blips) will remain eligible. Participant must have a complete antiretroviral treatment history including past and present data on resistance to antiretroviral therapy
4. Agree to continue their current antiretroviral regimen during the study period unless change in treatment with antiretroviral regimen is medically indicated
5. Have, in the Investigator's opinion, a fully active alternative antiretroviral regimen that can be used if resistance develops to the current antiretroviral therapy regimen
6. CD4 T cell count >400 cells/mm3
7. Has adequate organ function as indicated by the following laboratory values:

   * Hematocrit ≥33% or hemoglobin ≥13g/dL (males) and ≥12g/dL (females)
   * Platelet count ≥150,000/mm3
   * Absolute neutrophil count ≥1,500/mm3
   * Serum creatinine ≤1.3 times ULN or calculated creatinine clearance (for those with creatinine >1.3 ULN) ≥60mL/min
   * Prothrombin Time or INR ≤ 1.5 times ULN
   * Total bilirubin <1.5 times the ULN range. If total bilirubin is elevated, direct bilirubin must be < 2 times the ULN range, except in participants with Gilbert's Syndrome who must have serum bilirubin <3.0 times ULN (NOTE: If participant is on an atazanavir containing therapy then a direct bilirubin should be measured instead of the total bilirubin and must be ≤ 1.0mg/dL. Also, asymptomatic elevations due to ART medications are not exclusionary when, in the opinion of the Investigator, the abnormalities are not attributable to intrinsic hepatic disease).
   * Amylase < 3 times ULN at the time of screening
   * AST (SGOT) and ALT (SGPT): ≤ 3.0 times ULN
8. Adequate venous access, per Investigator judgement, and no other contraindications for leukapheresis
9. Weight (without shoes) ≥50 kilograms
10. Has the ability to understand the study and must be willing to comply with study-required procedures and visits
11. Written informed consent signed and dated by the study participant
12. A negative pregnancy test for females of childbearing potential. A female participant is considered to be of childbearing potential if she is menstruating, has an intact uterus and at least 1 ovary, and is less than 2 years postmenopausal.
13. Unless medically prescribed, a negative drug test for amphetamines; barbiturates; benzodiazepines; cocaine; methadone (Dolophine®); opiates (codeine, morphine only); phencyclidine (PCP); propoxyphene
14. Agree to participate in the 15-year Long-Term Follow-Up study

Exclusion Criteria:

1. Active viral hepatitis B or hepatitis C infection. A complete hepatitis B virus (HBV) screen (B-core antibody, HBV surface antibody, and HBV surface antigen testing) must be completed. Viral load testing will be used in questionable cases, per the discretion of the Investigator.

   * The results for hepatitis B may be positive for surface antibodies against HBV but must be negative for circulating HBV surface antigen to confirm the absence of active infection and negative for HBV core antigen to excluded previous active hepatitis
   * The results for hepatitis C virus (HCV) may be positive for antibodies against HCV but must be negative for HCV viral RNA in blood to confirm the absence of active infection.
2. Liver disease by any cause
3. Active or history (within 5 years prior to screening) of at least one acquired immune deficiency syndrome (AIDS)-defining complication
4. CD4 T cell nadir of <200 cells/mm3, if the information is available at the time of screening per medical records. If this information is unavailable, the Investigator will document this in the study source records
5. Cancer or malignancy that has not been in remission for at least 5 years prior to screening, with the exception of successfully treated basal cell carcinoma of the skin
6. Current diagnosis of congestive heart failure, uncontrolled angina, or arrhythmias
7. Baseline prolonged QTc (Fridericia Formula) of 450 ms or more
8. Any clinically significant renal, hepatic, or pulmonary disease
9. History of active or latent tuberculosis, regardless of treatment history
10. Asplenia
11. Received high dose cytoreduction therapy within 3 months prior to screening
12. Currently taking (or has taken within 6 months prior to screening) the antiretroviral drug Selzentry (Maraviroc)
13. Currently using protease inhibitors, efavirenz, or zidovudine
14. Prior events of hemorrhagic cystitis
15. Evidence of urinary outflow obstruction by history, enlarged prostate on physical exam, or use of medications for urinary outflow obstruction
16. Is being treated for culture-confirmed bacteremia or had culture-confirmed bacteremia within 1 month prior to screening
17. Has signs or symptoms of acute infectious disease
18. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
19. History of neurological diseases
20. Significant laboratory values and/or chronic medical condition that in the opinion of the Investigator could impact trial participation
21. Received another investigational drug or device within 30 days of screening
22. Previously received any gene transfer therapy
23. History or any features on physical examination indicative of a bleeding diathesis
24. Use of aspirin, dipyridamole, warfarin and antithrombin inhibitors or any other medication that is likely to affect platelet function or other aspects of blood coagulation within 3 days prior to the Leukapheresis Visit
25. Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., monoclonal antibodies, interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to screening (NOTE: Use of inhaled or topical steroids is not exclusionary)
26. Currently pregnant or breast-feeding
27. Unwilling to use acceptable methods of birth control for 6 months following the infusion of AGT103-T if sexually active with opposite sex. The following are acceptable methods of birth control: condoms (male or female) with or without a spermicidal agent, intrauterine device, diaphragm or cervical cap with spermicide, or hormonal-based contraception
28. Active alcohol use or dependence that, in the opinion of the Investigator, would interfere with adherence to study requirements
29. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to screening
30. Recent vaccination or intercurrent illness within 5 weeks prior to screening (NOTE: It is recommended that participants should have completed their routine vaccinations, e.g., hepatitis A or B, pneumococcus, influenza and tetanus diphtheria booster, at least 5 weeks prior to screening for the study)
31. Known allergy to Dimethyl Sulfoxide (DMSO)
32. Known allergy to Cyclophosphamide

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Assess the safety of AGT103-T in HIV+ participants with well-controlled viremia on antiretroviral therapy: adverse events | Days 1 to 180 post-infusion
  Incidence of adverse events related to AGT103-T will be graded using NCI CTCAE (v5.0)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Washington Health Institute, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jain A, Liou ML, Xiao L, Canepa GE. Impact of AGT103-T cell and gene therapy on intact HIV proviral reservoirs. AIDS. 2026 Feb 11. doi: 10.1097/QAD.0000000000004459. Online ahead of print. PMID 41670418
- [Derived] Pauza CD, Huang K, Bordon J. Advances in cell and gene therapy for HIV disease: it is good to be specific. Curr Opin HIV AIDS. 2021 Mar 1;16(2):83-87. doi: 10.1097/COH.0000000000000666. PMID 33625039